CLINICAL TRIAL: NCT07356713
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Trial of Exl-111 in Healthy Participants
Brief Title: A Study to Find a Suitable Dose of Exl-111 for Further Research
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Excellergy Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Exl-111.101
Record Dates: First submitted 2025-12-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Allergic Disease
MeSH Terms: interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exl-111 (SAD) (Experimental): Healthy participants receive a single subcutaneous dose of Exl-111 at 5 ascending dose levels
  Interventions: Drug: Exl-111 (SAD)
- Exl-111 (MAD) (Experimental): Healthy participants receive Exl-111 at 3 ascending dose levels administered every 4 weeks (Q4W) for a total of 4 doses
  Interventions: Drug: Exl-111 (MAD)
- Placebo (Experimental): Participants receive placebo injections matched in appearance and schedule to Exl-111: a single SC dose in Part A (SAD) or SC doses Q4W x4 in Part B (MAD), according to their assigned cohort.
  Interventions: Drug: Placebo
- Comparator (Experimental): (MAD) Healthy participants receive omalizumab injections every 4 weeks (Q4W) for a total of 4 doses
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Exl-111 (SAD) — Exl-111 is administered by subcutaneous injection in a single dose.
  Arms: Exl-111 (SAD)
Drug: Exl-111 (MAD) — Exl-111 is administered by subcutaneous injection in ascending dose levels.
  Arms: Exl-111 (MAD)
Drug: Placebo — A placebo matched in appearance and route of administration to Exl-111 is given by subcutaneous injection
  Arms: Placebo
Drug: Omalizumab — Omalizumab is administered by subcutaneous injection
  Arms: Comparator

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single and multiple ascending dose trial of Exl-111 in healthy participants.

The trials consists of 2 parts, as follows:

Part A (SAD): Up to 5 dose cohorts, each with 8 participants, randomized into 2 arms: Exl-111 and placebo.

Part B (MAD): Up to 3 dose cohorts, each with 10 participants, randomized into 3 arms: Exl-111, placebo, and an active comparator (omalizumab).

DETAILED DESCRIPTION:
Phase 1, randomized, double-blind, placebo-controlled, single and multiple ascending dose trial of Exl-111 in healthy participants.

Part A : In all SAD cohorts, trial intervention will be administered as single SC injection on Day 1. Participants will remain in the clinic through Day 5 and will return to the clinic for multiple follow up visits through Day 141 (Week 20)/End of Study [EOS]). The trial may proceed to Part B if recommended by the Safety Monitoring committee (SMC) upon review of available Part A safety data as described below.

Part B: Part B may be initiated following approval by the SMC after the SMC meeting for SAD Cohort 3 in Part A, and SMC review of:

SAD cohort corresponding to the proposed MAD starting dose level and SAD cohort corresponding to the proposed dose above the MAD starting dose level Participants will remain in the clinic from Day -1 through Day 5 for the first dose, Days 28-31 for the second dose, Days 56-59 for the third dose, and Days 84-89 for the fourth dose. Following the last dose, participants will return to the clinic over multiple follow-up assessments through Day 196 (Week 28)/EOS, 16 weeks after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male and female participants 18-55 years of age at Screening
2. Body weight ≥45 kg and ≤120 kg and body mass index (BMI) 18 to ≤32 kg/m2 at Screening and Day -1
3. Serum IgE ≥30 IU/mL and ≤300 IU/mL at Screening
4. Nonsmoker and must not have used any tobacco products within 2 months prior to Screening. Participants who smoke ≤2 cigarettes or equivalent (e.g., cigars, vaping, nicotine patches) per week can be included in the trial at the discretion of the PI/delegate
5. Positive skin prick test at Screening (Part B MAD Cohorts only) to common aeroallergens
6. Willing and able to read, understand, and sign an informed consent form (ICF) that includes compliance with requirements and restrictions listed in the ICF and in this protocol

Exclusion Criteria:

1. Received Exl-111 in a prior cohort in this trial
2. Prior receipt of any anti-IgE therapy
3. Use of any medication, including any prescription, over-the-counter, or other supplements, within 5 days prior to dosing, extending to 30 days after last dose of trial intervention, with the exception of those approved by the PI and Sponsor or Sponsor representative.
4. Receipt of any small molecule investigational agent or trial intervention in a clinical trial within 30 days or 5 half-lives (whichever is longer) prior to Day 1
5. Receipt of any protein or antibody-based therapeutic agents (e.g., growth hormones or mAbs) within 3 months or 5 half-lives (whichever is longer) prior to Screening
6. Receipt of either of the following:

   1. Any live/unattenuated vaccinations within 12 weeks prior to Screening
   2. Non-living/attenuated vaccinations (including inactivated vaccines, messenger RNA vaccines) within 4 weeks prior to Screening
7. History of active systemic infection within 30 days prior to Day 1
8. Known history of positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), human immunodeficiency virus (HIV)-1 or HIV-2
9. Positive test at Screening for HBsAg, hepatitis B core antibody (HBcAb), HCV Ab, HIV antibody, QuantiFERON®-TB Gold In-Tube test
10. Active treatment for any allergic condition, except for over-the-counter (OTC) antihistamines for seasonal allergy subject to exclusion #11
11. In Part B only, use of any drug that may interfere with the skin prick test results, including antihistamine use within 5 days before each skin prick test
12. History of relevant drug hypersensitivity, or any confirmed significant allergic reactions (urticaria or anaphylaxis), as judged by the PI, against any drug, or multiple drug or food allergies.
13. History of cardiac arrhythmia or family history of sudden cardiac death or a history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, hypomagnesia, or family history of Long QT Syndrome)
14. Clinically relevant history of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, endocrinological, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, ophthalmological, or connective tissue diseases or disorders that, in the opinion of the PI, might pose additional risk to the participant or confound the results of the trial
15. History of malignancy in the previous 5 years
16. History of alcohol or substance use disorder within the previous 5 years
17. History of vasovagal reactions
18. History of hereditary alpha-tryptasemia
19. Positive test result for alcohol or drugs of abuse at Screening or Day -1
20. Clinical laboratory safety test results outside the local reference range at Screening or Day -1 which are deemed to be clinically significant by PI/delegate
21. AST/ALT >1.5 × ULN or total bilirubin > ULN at Screening or Day -1 (excluding participants with documented history of Gilbert's syndrome)
22. Screening or Day -1 estimated glomerular filtration rate <60 mL/min/1.73m2, according to the Chronic Kidney Disease Epidemiology Collaboration equation. Borderline results (±10 mL/min/1.73m2) may be acceptable based on PI's discretion.
23. Screening or Day -1 supine blood pressure (BP) ≥160 mmHg (systolic) or ≥95 mmHg (diastolic), following at least 5 minutes of supine rest. If BP is ≥160 mmHg (systolic) or ≥95 mmHg (diastolic), the BP should be repeated 2 more times (at least 5 minutes between measures) and the average of the 3 BP values should be used to determine the participant's eligibility
24. Screening supine 12-lead ECG demonstrates a QTcF interval >450 msec for male participants or >470 msec for female participants, or a QRSD interval >120 msec or any other relevant ECG finding at Screening. If the QTcF exceeds 450 msec, or QRSD exceeds 120 msec, the ECG should be repeated 2 more times (at least 5 minutes between measures) and the average of the 3 QTcF or QRSD values should be used to determine the participant's eligibility
25. Pregnant, lactating, or breastfeeding, or plan to become pregnant while participating in the trial or within 30 days of the last dose of trial intervention
26. Unwilling or unable to comply with the contraception requirements and lifestyle restrictions
27. Employee of the Sponsor or the site or a relative of an employee at the site

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-12-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events and serious adverse events for Part A and Part B | From first dose through Day 196.
  This is to evaluate the safety and tolerability of single and multiple dose administration of Exl-111 in healthy participants

SECONDARY OUTCOMES:
Pharmacokinetic assessment of maximum observed plasma concentration (Cmax) of Exl-111 | From treatment Day 1 to EOS/ET Week 20.
  Maximum plasma concentration (Cmax)
Pharmacokinetic assessment of Time to Maximum Concentration (Tmax) of Exl-111 | From treatment Day 1 to EOS/ET Week 20.
  Time to Maximum Concentration (Tmax)
Pharmacokinetic assessment apparent Terminal Half-life (t1/2) of Exl-111 | From treatment Day 1 to EOS/ET Week 20.
  Terminal Half-life (t1/2)
Pharmacokinetic assessment observed volume of distribution associated with the terminal slope following administration of Exl-111. ( VZO) | From treatment Day 1 to EOS/ET Week 20.
  Volume of distribution ( VZO)
Pharmacokinetic assessment area under the curve (AUC) from the time of dosing to the last measurable concentration of Exl-111. (AUCLST) | From treatment Day 1 to EOS/ET Week 20.
  Area Under the Curve (AUC)
Pharmacokinetic assessment the area under the curve (AUC) extrapolated to infinity from dosing time, based on the last observed concentration of Exl-111. (AUCIFO) | From treatment Day 1 to EOS/ET Week 20.
  Area under the curve (AUC) based on the last observed concentration. (AUCIFO)
Pharmacokinetic assessment the area under the curve (AUC) extrapolated to t from dosing time, based on tau of Exl-111. (AUCT) | From treatment Day 1 to EOS/ET Week 20.
  Area Under the Curve Over the Dosing Interval (AUCT) Assessment
Pharmacokinetic assessment the maximum concentration occurring at Tmax, divided by the dose of Exl-111. (CMAXD) | From treatment Day 1 to EOS/ET Week 20.
  Dose-Normalized Maximum Plasma Concentration (Cmax/D)
Pharmacokinetic assessment the area under the curve (AUC) for the defined interval between doses (TAU) divided by the dose of Exl-111. (AUCTAUD) | From treatment Day 1 to EOS/ET Week 20.
  Pharmacokinetic assessment the area under the curve (AUC) for the defined interval Dose-Normalized Area Under the Curve Over the Dosing Interval (AUCTAUD)

IPD SHARING:
Plan to Share IPD: No